CLINICAL TRIAL: NCT01570634
Title: Proof-of-Concept, CASAD for Treatment of Clostridium Difficile Infection
Brief Title: Proof-of-Concept, Calcium Aluminosilicate Anti-Diarrheal (CASAD) for Treatment of Clostridium Difficile Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped for slow enrollment - only 2 patients, no evaluable results
Sponsor: Salient Pharmaceuticals Incorporated (Industry)
Collaborators: Scott and White Hospital & Clinic (Other); Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAL-2011-01PCL-01
Record Dates: First submitted 2012-04-01; First posted 2012-04-04 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Diarrhoea, Clostridium Difficile
Keywords: Clostridium difficile; infection; diarrhea; cramping
MeSH Terms: conditions — Diarrhea; Infections; Spasm | interventions — Calcium Aluminosilicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label CASAD (Experimental): Treatment with CASAD for 14 days
  Interventions: Drug: Calcium Aluminosilicate Anti-Diarrheal (CASAD)

INTERVENTIONS:
Drug: Calcium Aluminosilicate Anti-Diarrheal (CASAD) — CASAD 3 500mg capsules po tid for 14 days with 4 weeks of follow up
  Other Names: CASAD

SUMMARY:
Clostridium difficile (C. difficile) can cause symptoms ranging from mild diarrhea to life-threatening colitis. Illness from C. difficile most commonly affects patients in hospitals and long-term care facilities and typically occurs after a patient has received antibiotics.

In vitro data indicate Calcium Aluminosilicate Anti-Diarrheal (CASAD) has the potential to bind TNFα, IL-1, IL-6, and IL-10 in the intestines and, therefore, may act to reduce severity of fever, leukocytosis, and bowel injury in patients with C. difficile infection. This would likely occur in conjunction with neutralization of C. difficile toxins A&B by CASAD. Computer modeling of CASAD performed by Phillips et al. at Texas A&M University supports this hypothesis.

The investigators hypothesize that adding CASAD 1.5 grams po tid to any standard-of-care therapy will reduce the duration and severity of diarrhea and other symptoms in patients with C. difficile infection.

ELIGIBILITY:
Inclusion Criteria:

* C. difficile-associated diarrhea at the time of enrollment
* 18 years old and up
* Ability to take oral medications
* Negative urine pregnancy test for women of childbearing age
* Must have the ability to understand and the willingness to provide a written informed consent to participate in the study

Exclusion Criteria:

* History of known allergy to silicates
* Patients with signs of toxic megacolon, peritonitis, pseudomembranous colitis or bowel perforation
* Patients with hypotension (systolic blood pressure < 90 mm Hg) or septic shock requiring pressors
* Patients with other known causes of diarrhea or colitis
* Pregnancy or lactation
* History of significant neurological or psychiatric disorders that would impede giving consent, treatment, or follow up
* Participation in any other study where the subject is actively taking investigational medication within the last 30 days
* More than 5 doses of metronidazole or oral vancomycin prior to starting on study drug for the current C. difficile diagnosis. Administration of metronidazole or oral vancomycin for treatment of prior C. difficile diagnosis is not exclusionary as some patients may be experiencing a relapse of C. difficile.
* Any other antibiotic, toxin-binding agent or fecal transplant used for the treatment of C. difficile prior to or added to the subject's standard-of-care treatment regimen. Use of intravenous vancomycin is not exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarthi Narasimhan, MD, Principal Investigator — Scott & White Memorial Hospital
Locations (1):
- Scott & White Memorial Hospital, Temple, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting was managed by Scott & White
Groups:
- Open Label CASAD: Treatment with Calcium Aluminosilicate Anti-Diarrheal (CASAD) for 14 days
Period: Overall Study
Arm/Group | Open Label CASAD
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label CASAD
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 66.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Diarrhea
Description: To evaluate the safety and efficacy of CASAD added to the standard-of-care for the therapy of Clostridium difficile infection (C. difficile).
Time Frame: 42 days
Population: The study was terminated early due to slow enrollment. Of the 2 patients enrolled, one took less than 50% of the prescribed study drug. The results are not evaluable.
Arm/Group | Open Label CASAD
Number analyzed (Participants) | 0

2. Secondary Outcome: Stools Per Day
Description: Compare the number of liquid stools per day during treatment period
Time Frame: 14 days
Population: The study was terminated early due to slow enrollment. One of the two patients enrolled took less than 50% of the prescribed study drug.
Arm/Group | Open Label CASAD
Number analyzed (Participants) | 0

3. Secondary Outcome: Resolution of Abdominal Pain
Description: Compare time to resolution of abdominal pain
Time Frame: 14 days
Population: as for outcome 2
Arm/Group | Open Label CASAD
Number analyzed (Participants) | 0

4. Secondary Outcome: Absence of Relapse
Description: Compare sustained clinical response
Time Frame: 42 days
Population: as for outcome 2
Arm/Group | Open Label CASAD
Number analyzed (Participants) | 0

5. Secondary Outcome: Side-effects and Complications
Description: Compare side-effects and complications
Time Frame: 42 days
Population: as for outcome 2
Arm/Group | Open Label CASAD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during active study period of 6 weeks.
Arm/Group | Open Label CASAD
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label CASAD (N=2)
Nausea (Gastrointestinal disorders) | 1 (1) — unrelated to study drug, patient recovered with no residual effect.
Bloating (Gastrointestinal disorders) | 1 (1) — probably related to study drug, patient recovered, no action taken
Burping/Gas (Gastrointestinal disorders) | 1 (1) — Possible relationship to study drug, no action taken, patient recovered
Dark urine (Renal and urinary disorders) | 1 (1) — No action taken, patient recovered with no residual effects

LIMITATIONS AND CAVEATS:
This study was terminated early for slow enrollment. Only 2 patients were enrolled during the open period. One of the two took less than 50% of the prescribed study drug. The results are not meaningful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days